CLINICAL TRIAL: NCT03355911
Title: Relationship Between Preoperative Corneal Thickness and Postoperative
Brief Title: Preoperative Corneal Thickness and Postoperative Visual Outcomes After Posterior Lamellar Corneal Transplant
Acronym: TransCor
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-07Obs-CHRMT
Record Dates: First submitted 2017-11-23; First posted 2017-11-28 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Corneal Changes of Membranes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the impact of preoperative corneal thickness on visual outcomes following Descemet's stripping endothelial keratoplasty (DSAEK) or Descemet membrane endothelial keratoplasty (DMEK)

DETAILED DESCRIPTION:
Patients underwent DSAEK or DMEK for endothelial dysfunction, from October 2013 to November 2016. Patients aged > 18 years and with an indication for posterior lamellar graft surgery, such as Fuchs dystrophy, were included. Exclusion criteria included a history of penetrating keratoplasty in the study eye and a need for a penetrating keratoplasty following endothelial graft failure. Visual acuity, central corneal thickness (CCT) and graft thickness were measured preoperatively, and at postoperative day 7 and months 1, 3 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Clinically indicated need for posterior lamellar graft surgery (DSAEK or DMEK) such as:

  * Fuchs dystrophy,
  * pseudophakic bullous decompensation
  * or other endothelial dysfunction corneal

Exclusion Criteria:

* were a history of penetrating keratoplasty in the indicated eye
* the technical inability of preoperative CCT measurement
* the need for a penetrating keratoplasty following endothelial graft failure
* severe postoperative complications resulting in unquantifiable visual acuity

Age Groups: Child, Adult, Older Adult
Study Population: patients underwent posterior lamellar graft during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Descemet's stripping endothelial keratoplasty (DSAEK) or Descemet membrane endothelial keratoplasty (DMEK) | month 6
  LogMar

IPD SHARING:
Plan to Share IPD: Undecided